CLINICAL TRIAL: NCT00496327
Title: Evaluation of Safety,Tolerability and Immunogenicity of Vaccination With VARIVAX (V210)in Healthy Indian Children
Brief Title: Safety,Tolerability and Immunogenicity of Vaccination With VARIVAX in Healthy Indian Children (V210-056)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V210-056; 2007_019
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Herpes Zoster Vaccine

ARMS (1):
- 1 (Experimental): Open label
  Interventions: Biological: Varicella Virus Vaccine Live (Oka-Merck)

INTERVENTIONS:
Biological: Varicella Virus Vaccine Live (Oka-Merck) — VARIVAX(TM) (Refrigerated) [Varicella Virus Vaccine Live (Oka/Merck), Refrigerator-Stable Formulation.] Subjects enrolled in the study received one 0.5 mL subcutaneous dose of VARIVAX(TM). Frequency is single dose.

SUMMARY:
To observe the safety and tolerability of the administration of VARIVAX in varicella history negative Indian children 12 months to 12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children, Between 12 Months And 12 Years Of Age
* Parent Or Legal Guardian Should Be Willing And Able To Sign The Informed Consent Form Prior To Entry Into The Study

Exclusion Criteria:

* Any Immune Impairment Or Deficiency, Neoplastic Disease, Or Depressed Immunity, Including That Resulting From Corticosteroid Or Other Immunosuppressive Therapy
* Any Immunoglobulin Or Blood Products 5 Months Prior To Or Expected Within 3 Months After Enrollment In This Study

Any Medical Condition Which, In The Opinion Of The Investigator May Interfere With The Evaluation Of Teh Study Objectives

* Any Other Inactivated Vaccine Administered Within 14 Days Before Or Expected Within 42 Days After Administration Of The Study Vaccination
* Any Other Live Vaccine Administered Within 30 Days Before Or Expected Within 42 Days After Administration Of The Study Vaccination
* Female Subjects Who Are Pregnant Or Nursing
* History Of Anaphylactic Or Other Immediate Allergic Reactions
* Hypersensitivity To Any Of The Components Of The Vaccine Administered Under This Protocol Such As Gelatin Or Neomycin
* Past History Of Varicella
* Previous Vaccination With Any Varicella Vaccine In Either Monovalent Or Combination Form
* Recent Household, Daycare, Or School Exposure(In The Last 4 Weeks) To Varicella

Ages: 12 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2005-06-22 (Actual); Primary Completion 2005-10-06 (Actual); Study Completion 2005-10-06 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with VZV specific antibody titre>= 5gp ELISA units/ml 6 weeks post-vaccination | 6 weeks post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Subba Rao SD, Panday S, Maiya PP, Samdani PG, Lokeshwar MR, Bhave S, Bafna S. Immunogenecity and safety of Oka varicella-zoster virus vaccine (VaripedTM) in Indian children. New Indian Journal of Pediatrics. 2018;7.1(Jan-Mar):7-14. https://nijp.org/immunogenicity-and-safety-of-oka-varicella-zoster-virus-vaccine-varipedtm-in-indian-children/
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html